CLINICAL TRIAL: NCT04276688
Title: An Open-label Randomized Controlled Trial on Lopinavir/ Ritonavir, Ribavirin and Interferon Beta 1b Combination Versus Lopinavir/ Ritonavir Alone, as Treatment for 2019 Novel Coronavirus Infection
Brief Title: Lopinavir/ Ritonavir, Ribavirin and IFN-beta Combination for nCoV Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Hospital Authority, Hong Kong (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UW-20-074
Record Dates: First submitted 2020-02-11; First posted 2020-02-19 (Actual); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Novel Coronavirus Infection
Keywords: nCoV; lopinavir/ ritonavir; IFN-beta
MeSH Terms: interventions — Lopinavir; Ribavirin; Interferon beta-1b

STUDY DESIGN:
Intervention Model Description: open-label randomised controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Active Comparator): triple combination
  Interventions: Drug: Lopinavir/ritonavir; Drug: Ribavirin; Drug: Interferon Beta-1B
- Control group (Active Comparator): single
  Interventions: Drug: Lopinavir/ritonavir

INTERVENTIONS:
Drug: Lopinavir/ritonavir — 400mg/100mg twice daily for 14 days
Drug: Ribavirin — 400mg twice daily for 14 days
  Arms: Study group
Drug: Interferon Beta-1B — 0.25mg subcutaneous injection alternate day for 3 days
  Arms: Study group

SUMMARY:
A combination of lopinavir/ ritonavir, ribavirin and interferon beta-1b will expedite the recovery, suppress the viral load, shorten hospitalisation and reduce mortality in patients with 2019-n-CoV infection compared with to lopinavir/ ritonavir

DETAILED DESCRIPTION:
Hypothesis A combination of lopinavir/ ritonavir, ribavirin and interferon beta-1b will expedite the recovery, suppress the viral load, shorten hospitalisation and reduce mortality in patients with 2019-n-CoV infection compared with to lopinavir/ ritonavir alone

Primary objective: To evaluate the safety and efficacy in mortality reduction with a combination of lopinavir/ ritonavir, ribavirin and interferon beta-1b in the treatment of patient hospitalised for 2019-n-CoV infection and compare this to lopinavir/ ritonavir alone

Subject/patient definition: Recruited subjects include adult patients ≥18 years of age, admitted to the HA Hospitals from February 2020 onwards, with laboratory confirmed 2019-n-CoV infection. All subjects give written informed consent. Subjects must be available to complete the study and comply with study procedures.

Study design: This is a prospective open-label randomised controlled trial among adult patients hospitalised after February 2020 for virologically confirmed 2019-n-CoV infection. Patients will be randomly assigned to either a 14-day course of lopinavir/ ritonavir 400mg/100mg twice daily, ribavirin 400mg bd and zero to three doses of subcutaneous injection of interferon beta-1b 1mL (0.25mg; 8 million IU) on day 1, 3 and 5 (depending on day of admission from symptoms onset) plus standard care, or a 14-day course of lopinavir/ ritonavir 400mg/100mg twice daily plus standard care alone (2:1).

Intervention/study article: lopinavir/ ritonavir, ribavirin and interferon beta-1b

Primary outcome: Time to negative nasopharyngeal swab (NPS) 2019-n-CoV coronavirus viral RT-PCR

Secondary outcome:

1. Time to negative saliva 2019-n-CoV coronavirus viral RT-PCR
2. Time to clinical improvement of NEWS2 (National Early Warning Score 2) of 0 maintained for 24 hours
3. Length of hospitalisation
4. Adverse events during treatment
5. 30-day mortality
6. Cytokine/ chemokine changes

ELIGIBILITY:
Inclusion Criteria:

1. Recruited subjects include all adult patients ≥18 years hospitalised for virologically confirmed 2019-n-CoV infection.
2. NEWS of ≥1 upon recruitment
3. Auditory temperature ≥38°C with at least one of the following symptoms (cough, sputum production, sore-throat, nasal discharge, myalgia, headache or fatigue) upon admission
4. Symptom duration ≤10 days
5. All subjects give written informed consent.
6. Subjects must be available to complete the study and comply with study procedures. Willingness to allow for serum samples to be stored beyond the study period, for potential additional future testing to better characterize immune response.

Exclusion Criteria:

1. Inability to comprehend and to follow all required study procedures.
2. Allergy or severe reactions to the study drugs
3. Patients with known prolonged QT or PR interval, second- or third-degree heart block, or ventricular cardiac arrhythmias, including torsade de pointes
4. Patients taking medication that will potentially interact with lopinavir/ ritonavir, ribavirin or interferon-beta1b
5. Patients with known history of severe depression
6. Pregnant or lactation women
7. Inability to comprehend and to follow all required study procedures
8. Received an experimental agent (vaccine, drug, biologic, device, blood product, or medication) within 1 month prior to recruitment in this study or expect to receive an experimental agent during this study. Unwilling to refuse participation in another clinical study through the end of this study.
9. Have a history of alcohol or drug abuse in the last 5 years.
10. Have any condition that the investigator believes may interfere with successful completion of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2020-02-10 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Time to negative NPS | Up to 1 month
  Time to negative NPS 2019-n-CoV RT-PCR

SECONDARY OUTCOMES:
Time to negative saliva | Up to 1 month
  Time to negative saliva 2019-n-CoV RT-PCR
Time to clinical improvement | Up to 1 month
  Time to NEWS of 0
Hospitalisation | Up to 1 month
  Length of hospitalisation
Mortality | Up to 1 month
  30-day mortality
Immune reaction | up to 1 month
  Cytokine/ chemokine changes
Adverse events | up to 1 month
  Adverse events during treatment
Time to negative all clinical specimens | up to 1 month
  Time to negative NPS, saliva, urine and stool 2019-n-CoV RT-PCR

CONTACTS AND LOCATIONS:
Overall Officials: Ivan FN Hung, MD FRCP, Principal Investigator — The University of Hong Kong
Locations (1):
- University of Hong Kong, Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moschen AR. IBD in the time of corona - vigilance for immune-mediated diseases. Nat Rev Gastroenterol Hepatol. 2020 Sep;17(9):529-530. doi: 10.1038/s41575-020-0333-5. PMID 32555385
- [Derived] Hung IF, Lung KC, Tso EY, Liu R, Chung TW, Chu MY, Ng YY, Lo J, Chan J, Tam AR, Shum HP, Chan V, Wu AK, Sin KM, Leung WS, Law WL, Lung DC, Sin S, Yeung P, Yip CC, Zhang RR, Fung AY, Yan EY, Leung KH, Ip JD, Chu AW, Chan WM, Ng AC, Lee R, Fung K, Yeung A, Wu TC, Chan JW, Yan WW, Chan WM, Chan JF, Lie AK, Tsang OT, Cheng VC, Que TL, Lau CS, Chan KH, To KK, Yuen KY. Triple combination of interferon beta-1b, lopinavir-ritonavir, and ribavirin in the treatment of patients admitted to hospital with COVID-19: an open-label, randomised, phase 2 trial. Lancet. 2020 May 30;395(10238):1695-1704. doi: 10.1016/S0140-6736(20)31042-4. Epub 2020 May 10. PMID 32401715